CLINICAL TRIAL: NCT00203463
Title: Topiramate in the Treatment of Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuscaloosa Research & Education Advancement Corporation (Other)
Collaborators: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TREAC Topiramate in PTSD; TREAC Topiramate in PTSD
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-07-29 (Estimated); Status verified 2009-07

CONDITIONS: PTSD
Keywords: topiramate; PTSD; posttraumatic stress disorder; topamax
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
To study the potential therapeutic effects of topiramate (Topamax) in the treatment of PTSD.

DETAILED DESCRIPTION:
This is a twelve-week randomized, double blind, placebo controlled trial of topiramate for 40 patients with PTSD. Diagnoses are made by Structured Clinical Interview for DSM-IV (SCID). Symptom severity is measured with the Clinician Administered PTSD Scale (CAPS), Davidson Trauma Scale (DTS), Treatment Outcome PTSD (TOP-8), Clinical Global Impressions (CGI), and the Hamilton Rating Scales for Depression and Anxiety (HAM-D and HAM-A). The Clinician Administered PTSD Scale (CAPS) is the primary outcome measure. Subjects will read and sign informed consent prior to beginning any study procedures. Subjects who meet inclusion/exclusion criteria will be randomized 1:1 (Topiramate : placebo) to study medication. Study medication is initiated at one tablet daily (25mg topiramate or placebo) and medication will be increased by 25-100mg (1 tablet) increments every 7 days, as tolerated, until a maximum benefit is achieved, not to exceed 400mg/day. Patients will be seen every week up until Visit 4, and then will be seen every two weeks for the remainder of the study for assessment of efficacy and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD DSM-IV criteria
* No substance abuse/dependence for the previous 2 months (except for nicotine and caffeine)
* Free of psychotropic medication, for 2 weeks (except 6 weeks for fluoxetine)
* Normal physical and laboratory examination (lab profile listed below)
* Negative urine screen for drugs of abuse
* Women of childbearing potential must be using nonpharmacologic medically approved methods of birth control
* Signed informed consent
* Male or female, any race or ethic origin

Exclusion Criteria:

* Lifetime history of bipolar, psychotic, or cognitive disorders
* Suicidal, homicidal, or psychotic
* Diagnosis of bulimia or anorexia nervosa
* History of sensitivity to topiramate
* General medical conditions or ongoing treatment that contraindicate the use of topiramate, such as seizure disorder or use of MAO inhibitors.
* Women planning to become pregnant or breastfeed during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-07; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Potential therapeutic effects of topiramate (Topamax) in the treatment of PTSD as noted in the change of the 17-item total severity score of the Clinician-Administered PTSD scale (CAPS) from baseline to the last visit of Double-Blind Phase (8-weeks) | (8-weeks)

SECONDARY OUTCOMES:
Changes from baseline to the last visit in Double-Blind Phase for HAM-A, MADRS, and TOP-8 Scale, Clinical Global Impression (CGI)scales, and Davidson Trauma Scale (DTS). Each scale will be analyzed as described above for the primary efficacy variable. | (8-weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Lori L Davis, MD, Principal Investigator — Tuscaloosa Veterans Affairs Medical Center
Locations (1):
- Tuscaloosa Research & Education Advancement Corporation, Tuscaloosa, Alabama, United States

REFERENCES:
- [Background] Berlant JL. Topiramate in posttraumatic stress disorder: preliminary clinical observations. J Clin Psychiatry. 2001;62 Suppl 17:60-3. PMID 11495099